CLINICAL TRIAL: NCT02257138
Title: Phase I/II Study of Ruxolitinib Plus Decitabine in Patients With Post Myeloproliferative Neoplasm - Acute Myeloid Leukemia (AML)
Brief Title: Ruxolitinib Phosphate and Decitabine in Treating Patients With Relapsed or Refractory or Post Myeloproliferative Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0344; NCI-2014-02299 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0344 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-09-26; First posted 2014-10-06 (Estimated); Results first posted 2022-08-15 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Blasts More Than 20 Percent of Bone Marrow Nucleated Cells; Blasts More Than 20 Percent of Peripheral Blood White Cells; Myelodysplastic/Myeloproliferative Neoplasm; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute | interventions — Decitabine; Injections; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (ruxolitinib phosphate, decitabine) Ph1 (Experimental): Patients receive ruxolitinib phosphate PO BID on days 1-28 and decitabine IV on days 1-5. Treatment repeats every 4-6 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Other: Laboratory Biomarker Analysis; Drug: Ruxolitinib Phosphate
- Treatment (ruxolitinib phosphate, decitabine) Ph2 (Experimental): Patients receive 50mg ruxolitinib phosphate PO BID on days 1-28 and decitabine IV on days 1-5. Treatment repeats every 4-6 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Other: Laboratory Biomarker Analysis; Drug: Ruxolitinib Phosphate

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Aza-TdC; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi

SUMMARY:
This phase I/II trial studies the side effects and best dose of ruxolitinib phosphate when given together with decitabine and to see how well they work in treating patients with acute myeloid leukemia that has come back or is not responding to treatment, or has developed from a type of bone marrow diseases called myeloproliferative neoplasms. Ruxolitinib phosphate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ruxolitinib phosphate together with decitabine may be an effective treatment for acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the tolerability of the combination of decitabine and ruxolitinib phosphate (ruxolitinib [DI]) in patients with leukemia. (Phase I) II. To determine the efficacy of ruxolitinib in increasing and prolonging response induced by decitabine alone in patients with post myeloproliferative neoplasm acute myeloid leukemia (AML) (post MPN-AML) alternatively referred to as (myeloproliferative neoplasm - blast phase; MPN-BP). (Compared to historical response rate with decitabine alone) (Phase II)

SECONDARY OBJECTIVES:

I. To compare whether there is a difference in response rate patients with post-MPN AML with janus kinase 2 (JAK2) mutations and patients without JAK2 mutations.

OUTLINE: This is a phase I, dose-escalation study of ruxolitinib phosphate followed by a phase II study.

Patients receive ruxolitinib phosphate orally (PO) twice daily (BID) on days 1-28 and decitabine intravenously (IV) over 1-2 hours on days 1-5. Treatment repeats every 4-6 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML (World Health Organization [WHO] classification definition of >= to 20% blasts)
* In the phase I portion of the study all patients with relapsed or refractory AML are eligible; for the Phase II portion of the study, patients must have AML progressing from prior MPN (MPN-BP) or have myelodysplastic syndrome (MDS)/MPN with more than 20% blasts; temporary prior measures to control blood counts, such as apheresis or Hydrea are allowed; patients with newly diagnosed or previously treated disease are eligible as long as prior therapy does not include hypomethylating agents; prior therapy for ruxolitinib for MPN is allowed
* Serum biochemical values with the following limits unless considered due to leukemia:
* Creatinine =< 1.5 mg/dl
* Total bilirubin =< 1.5 mg/dL, unless increase is due to hemolysis or congenital disorder
* Transaminases (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x upper limit of normal (ULN)
* Ability to take oral medication
* Ability to understand and provide signed informed consent
* Performance status =< 3, unless directly related to disease process as determined by the principal investigator

Exclusion Criteria:

* Any coexisting medical condition that in the judgment of the treating physician is likely to interfere with study procedures or results including uncontrolled severe infections, as well as uncontrolled cardiac disease, or other organ dysfunction; patients with history of tuberculosis, human immunodeficiency virus (HIV) or hepatitis B and C are excluded
* Nursing women, women of childbearing potential with positive blood pregnancy test within 30 days of study start, or women of childbearing potential who are not willing to maintain adequate contraception (such as birth control pills, intrauterine device [IUD], diaphragm, abstinence, or condoms by their partner) over the entire course of the study
* Incomplete recovery from any prior surgical procedures or had surgery within 4 weeks prior to study entry, excluding the placement of vascular access
* Active clinically serious and uncontrolled infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment Period: February 2015 to March 2021
Groups:
- Ph1 (MTD) 10mg; Ph1 (MTD) 15mg; Ph1 (MTD) 25mg; Ph1 (MTD) 50mg; Ph2 Treatment (Ruxolitinib Phosphate, Decitabine): Patients receive ruxolitinib phosphate PO BID on days 1-28 and decitabine IV on days 1-5. Treatment repeats every 4-6 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Decitabine: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Ruxolitinib Phosphate: Given PO
Period: Overall Study
Arm/Group | Ph1 (MTD) 10mg | Ph1 (MTD) 15mg | Ph1 (MTD) 25mg | Ph1 (MTD) 50mg | Ph2 Treatment (Ruxolitinib Phosphate, Decitabine)
Started | 5 | 3 | 3 | 3 | 16
Completed | 5 | 3 | 3 | 3 | 16
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ph2 Treatment (Ruxolitinib Phosphate, Decitabine): Patients receive 50mg ruxolitinib phosphate PO BID on days 1-28 and 20mg/m^2 decitabine IV on days 1-5. Treatment repeats every 4-6 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Decitabine: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Ruxolitinib Phosphate: Given PO
- Total: Total of all reporting groups
Arm/Group | Ph1 (MTD) 10mg | Ph1 (MTD) 15mg | Ph1 (MTD) 25mg | Ph1 (MTD) 50mg | Ph2 Treatment (Ruxolitinib Phosphate, Decitabine) | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 2 | 7 | 11
  >=65 years | 4 | 3 | 2 | 1 | 9 | 19
Age, Continuous [Median (Full Range); unit: years] | 84 [32 to 92] | 69 [68 to 80] | 77 [65 to 80] | 61 [54 to 71] | 69 [46 to 79] | 69 [32 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 0 | 6 | 11
  Male | 2 | 2 | 2 | 3 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 3 | 4
  White | 5 | 3 | 2 | 3 | 10 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 3 | 3 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Ruxolitinib Phosphate (Phase I)
Description: Maximum tolerated dose (MTD) is defined as the highest dose studied for which the incidence of dose-limiting toxicity (DLT) is less than or equal to 17% (1 out of 6).
Time Frame: Up to 6 weeks
Measure: Number; unit: Dose in Milligrams
Groups:
- Ph1 (MTD) Treatment (Ruxolitinib Phosphate, Decitabine): Patients receive ruxolitinib phosphate PO BID on days 1-28 and decitabine IV on days 1-5. Treatment repeats every 4-6 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Decitabine: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Ruxolitinib Phosphate: Given PO
Arm/Group | Ph1 (MTD) Treatment (Ruxolitinib Phosphate, Decitabine)
Number analyzed (Participants) | 14
Dose in Milligrams | NA — Maximum Tolerated Dose (MTD) was not reached in this study as there were no Dose Limiting Toxicities (DLT) as defined in the Outcome Measure Description. The highest dose in the phase 1 portion of this study was 50 milligrams (mg) of ruxolitinib. The study continued to phase 2, treating all participants with 50mg ruxolitinib.

2. Primary Outcome: Number of Participants With a Response (Complete Response [CR] + CR With Incomplete Blood Count Recovery) (Phase 2)
Description: Complete Response (CR) is defined as - The participant must be free of all symptoms related to leukemia and have an absolute neutrophil count >/= 1 z 10^9/L, no need for red blood cell transfusion, platelet count>/+ 100 x 10^9/L, and normal marrow differential (</= 5 % blasts) in a normo- or hypercellular marrow. Complete Response with incomplete blood count recovery (CRi) is defined as - Same as CR but incomplete count recovery.
Time Frame: Up to 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ph2 Treatment (Ruxolitinib Phosphate, Decitabine)
Number analyzed (Participants) | 16
Participants | 8

3. Primary Outcome: Number of Participants With Post-MPN Acute Myeloid Leukemia (AML) With JAK2 Mutations (Phase 2)
Description: JAK2 mutations were assessed with the baseline Bone Marrow or Peripheral Blood.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Ph2 Treatment (Ruxolitinib Phosphate, Decitabine)
Number analyzed (Participants) | 16
Participants | 11

4. Secondary Outcome: Number of JAK2 Positive+ and JAK2 Negative- Participants With a Response (Phase 2)
Description: JAK2 mutations were assessed with the baseline Bone Marrow or Peripheral Blood. Complete Response (CR) is defined as - The participant must be free of all symptoms related to leukemia and have an absolute neutrophil count >/= 1 z 10^9/L, no need for red blood cell transfusion, platelet count>/+ 100 x 10^9/L, and normal marrow differential (</= 5 % blasts) in a normo- or hypercellular marrow. Complete Response with incomplete blood count recovery (CRi) is defined as - Same as CR but incomplete count recovery.
Time Frame: up to 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ph2 Treatment (Ruxolitinib Phosphate, Decitabine)
Number analyzed (Participants) | 8
Participants
  JAK 2+ Positive | 5
  JAK 2- negative | 3

ADVERSE EVENTS:
Time Frame: Up to 6 years
Arm/Group | Ph1 (MTD) 10mg | Ph1 (MTD) 15mg | Ph1 (MTD) 25mg | Ph1 (MTD) 50mg | Ph2 Treatment (Ruxolitinib Phosphate, Decitabine)
All-Cause Mortality (participants affected / at risk) | 2/5 | 3/3 | 1/3 | 2/3 | 2/16
Serious Adverse Events (participants affected / at risk) | 3/5 | 3/3 | 3/3 | 3/3 | 11/16
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 3/3 | 3/3 | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph1 (MTD) 10mg (N=5) | Ph1 (MTD) 15mg (N=3) | Ph1 (MTD) 25mg (N=3) | Ph1 (MTD) 50mg (N=3) | Ph2 Treatment (Ruxolitinib Phosphate, Decitabine) (N=16)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (5)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 2 (3) | 2 (4) | 3 (3) | 0 (0) | 5 (9)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lower Extremity Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph1 (MTD) 10mg (N=5) | Ph1 (MTD) 15mg (N=3) | Ph1 (MTD) 25mg (N=3) | Ph1 (MTD) 50mg (N=3) | Ph2 Treatment (Ruxolitinib Phosphate, Decitabine) (N=16)
Alkaline Phosphatase (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Elevated Bilirubin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Arrythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Elevated Creatinine (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema Limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage Gastrointestial (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage Other (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (3) | 2 (2)
Petechiae (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal/Genitourinary Other (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT02257138/Prot_SAP_000.pdf